CLINICAL TRIAL: NCT00654615
Title: The Fixation of Unstable Metaphyseal Distal Radius Fractures: A Randomized, Controlled Trial
Brief Title: Fixation of Unstable Distal Radius Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University (Other)
Collaborators: Stryker Trauma and Extremities (Industry)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00003715; GTS#32801 (Other: Wake Forest University Health Sciences)
Record Dates: First submitted 2008-04-02; First posted 2008-04-08 (Estimated); Results first posted 2017-11-13 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-08

CONDITIONS: Distal Radius Fractures
Keywords: unstable metaphyseal distal radius fractures; randomized controlled trial; surgical fixation; volar plate; intramedullary distal radius fixation system
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Intervention Model Description: This study was a prospective clinical trial comparing two different types of hardware to fix a specific type of distal radius fracture.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- 1 (Active Comparator): Intramedullary Radius Fixation (Micronail) - Group 1
  A new device was developed to provide intramedullary distal radius fracture fixation. This new device allows the placement of the orthopaedic hardware inside the medullary canal of the radius.
  Interventions: Device: Intramedullary Radius Fixation (Micronail)
- 2 (Active Comparator): Volar Plate Fixation - Group 2
  Volar locking plates provide rigid external fixation and are placed on the outside of the radius. Volar plates are placed directly on the distal radius using a metal plate contoured to the shape of the distal radius.
  Interventions: Procedure: Volar Plate Fixation

INTERVENTIONS:
Device: Intramedullary Radius Fixation (Micronail) — After adequate anesthesia was obtained and the patient was prepared for surgery, distraction was applied to the fracture site and preliminary reduction of the distal radius fracture was performed under fluoroscopic guidance. A pin was inserted to maintain the fracture reduction, then the Micronail was inserted inside the radius. The metaphyseal defect created by the fracture was filled using allograft or autograft bone material. Limited incisions at either the radial or ulnar columns was performed to achieve acceptable reduction of the fracture. Radiographic parameters were used to evaluate the results of the surgical management with intramedullary nailing.
  Arms: 1
Procedure: Volar Plate Fixation — After adequate anesthesia, longitudinal traction of the wrist was applied. Based on the fracture pattern, fragments were reduced and stabilized using either one 2.4mm titanium pre-contoured locking plate or a combination of locking plates. Arthrotomy was performed to verify that the fracture fragments were reduced. Plates were contoured to fit boney contours as needed. Allograft or autograft was placed in the fracture repair site as necessary. Radiographic landmarks were evaluated. Care was taken to ensure that plates were covered with periosteum or retinaculum to reduce the incidence of possible soft tissue irritation caused by the plate on the bone. The skin incision was closed; a removable splint applied.
  Arms: 2

SUMMARY:
Wrist fractures are the most common type of fractures that occur in the shoulder, arm, and hand. Approximately 250,000 to 300,000 wrist fractures occur in the United States each year. Although some wrist fractures can be treated using casts, many other fractures must be treated with surgery. The surgery involves using metal plates and screws to put the broken pieces of bone together so that they can heal. The purpose of this study is to compare two specific types of surgery that are used to treat broken wrists. One type uses pieces of metal that are placed on the outside of the broken pieces of bone that are screwed in place while the broken bones heal. The other type of surgery involves placing a piece of metal inside the bone marrow to hold the broken pieces of bone together as they heal. Individuals with broken wrists who participate in this study will be randomly assigned to receive one of the two types of surgical treatment. Both surgical treatments are approved and are not experimental. Study participants will be followed closely after surgery to determine the time required for them to return to their usual daily activities involving the use of their arms and hands. Although both groups of study participants are expected to experience the same outcomes at one year, those participants that receive the device placed inside the bone marrow may return to their normal functional activities earlier than the ones treated with the plate placed on the outside of the bone. Study participants and their surgeons will complete data sheets and questionnaires that will document their progress following treatment of their wrist fractures.

DETAILED DESCRIPTION:
INTRODUCTION: Fractures of the distal radius are the most common upper extremity fractures, accounting for approximately 250,000 to 300,000 injuries in the United States annually. The goals of treatment for patients with distal radius fractures are restoration of wrist anatomy, return of normal pain-free hand and wrist range of motion, and early return to normal activities of daily living. Management of distal radius fractures is dictated by the fracture pattern, the degree of displacement of the bone fragments, whether or not the fracture involves the joint, the presence of other bodily injuries, and the patient's pre-injury activity level and physical demands.

Unstable distal radius fractures require surgical fixation of the broken bone because closed reduction (nonsurgical manipulation of the fractured bones and casting) often is not sufficient to maintain fracture reduction and promote bone healing. Operative management of distal radius fractures has been studied extensively and has evolved over the past decade.

STUDY HYPOTHESIS: There are no published prospective, randomized trials comparing open reduction using volar plating to intramedullary fixation for the management of displaced unstable, metaphyseal distal radius fractures. The study hypothesis is that the outcomes of treatment of distal radius fractures using an intramedullary radius fixation system (Micronail®) will result in the earlier return of wrist range of motion, earlier functional recovery, and improvements in health-related quality of life equal to or superior to the outcomes of volar plate fixation.

SPECIFIC AIMS: The specific aim of this randomized, controlled clinical trial is to compare an intramedullary radius fixation system (Micronail®) to a volar locking plate technique for the management of displaced, unstable, metaphyseal distal radius fractures. Both functional and health-related quality of life outcomes of the study participants will be documented during the trial. In addition, radiographic information will be collected to compare the radiographic evidence of fracture healing in the two treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for participation in this study will include skeletally mature individuals between the ages of 18 through 80 who have sustained closed, displaced, unstable, metaphyseal fractures of the distal radius requiring surgical fixation.

Exclusion Criteria:

* Patients ineligible for study participation will include:

  * patients with multitrauma who must be treated in the ICU for long periods of time
  * patients with open wrist fractures,
  * patients who are skeletally immature,
  * patients with concomitant scaphoid fractures or other hand injuries that impact functional recovery,
  * patients with bilateral arm fractures or comminuted intraarticular distal radius fractures,
  * patients who have sustained previous wrist injury of the affected arm,
  * signs of rheumatoid arthritis, osteoarthritis, or polyarthritis, and
  * patients with physical or mental issues that make obtaining informed consent impossible.
* Any comorbid health conditions of the study participants (e.g. high blood pressure, COPD) will be documented.
* Patients who are interested in participating in this study will be asked to provide informed consent prior to their entry into the study protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-05; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zhongyu Li, MD, PhD, Principal Investigator — Assistant Professor
Locations (1):
- Wake Forest University Health Sciences - CompRehab, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Intramedullary Radius Fixation (Micronail) - Group 1: Intramedullary Radius Fixation (Micronail) - Group 1
  A new device was developed to provide intramedullary distal radius fracture fixation. This new device allows the placement of the orthopaedic hardware inside the medullary canal of the radius.
  Intramedullary Radius Fixation (Micronail): After adequate anesthesia was obtained and the patient was prepared for surgery, distraction was applied to the fracture site and preliminary reduction of the distal radius fracture was performed under fluoroscopic guidance. A pin was inserted to maintain the fracture reduction, then the Micronail was inserted inside the radius. The metaphyseal defect created by the fracture was filled using allograft or autograft bone material. Limited incisions at either the radial or ulnar columns was performed to achieve acceptable reduction of the fracture. Radiographic parameters were used to evaluate the results of the surgical management with intramedullary nailing.
- Volar Plate Fixation - Group 2: Volar Plate Fixation - Group 2
  Volar locking plates provide rigid external fixation and are placed on the outside of the radius. Volar plates are placed directly on the distal radius using a metal plate contoured to the shape of the distal radius.
  Volar Plate Fixation: After adequate anesthesia, longitudinal traction of the wrist was applied. Based on the fracture pattern, fragments were reduced and stabilized using either one 2.4mm titanium pre-contoured locking plate or a combination of locking plates. Arthrotomy was performed to verify that the fracture fragments were reduced. Plates were contoured to fit boney contours as needed. Allograft or autograft was placed in the fracture repair site as necessary. Radiographic landmarks were evaluated. Care was taken to ensure that plates were covered with periosteum or retinaculum to reduce the incidence of possible soft tissue irritation caused by the plate on the bone. The skin incision was closed; a removable splint applied.
Period: Overall Study
Arm/Group | Intramedullary Radius Fixation (Micronail) - Group 1 | Volar Plate Fixation - Group 2
Started | 30 | 30
Completed | 22 | 23
Not Completed | 8 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intramedullary Radius Fixation (Micronail) - Group 1 | Volar Plate Fixation - Group 2 | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 23 | 47
  >=65 years | 6 | 7 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] — Participants between the ages of 18 and 80 were enrolled.
  years | 55 (14) | 55 (16) | 55 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 19 | 44
  Male | 5 | 11 | 16
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Average Difference Between Michigan Hand Outcomes Questionnaire Scores
Description: Developed at the University of Michigan Department of Plastic Surgery to evaluate outcomes and function in patients who sustain upper extremity injuries. This will be done one week post-surgery compared to six weeks post-surgery comparing the two groups. The MHQ contains six domains: overall hand function, activities of daily living, work performance, pain, aesthetics, satisfaction. In the pain scale, high scores indicate greater pain, while in the other five scales, high scores denote better hand performance. The raw scale score for each of the six scales is the sum of the responses of each scale item. The raw score is converted to a score ranging from 0-100. An overall MHQ score can be obtained by summing the scores for all six scales after reversing the pain scale (pain=100-pain score) and then dividing by six. The overall MHQ score ranged between 0-100. Higher scores indicate better hand performance.
Time Frame: two week post-surgery compared to six weeks post-surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intramedullary Radius Fixation (Micronail) - Group 1 | Volar Plate Fixation - Group 2
Number analyzed (Participants) | 30 | 30
units on a scale | 85.2 (6.5) | 91.8 (4.2)

2. Secondary Outcome: Disabilities of the Arm, Shoulder, and Hand Questionnaire (DASH)
Description: The Disabilities of the Arm, Shoulder, and Hand Questionnaire (DASH) is a 30-item, self-report questionnaire designed to measure physical function and symptoms in patients with any or several musculoskeletal disorders of the upper limb. Each question is scored 1-5 with 1 meaning the least amount of severity of pain or difficulty and 5 meaning the maximum amount of pain or difficulty possible. At least 27 of the 30 items must be completed for a score to be calculate. All responses are summed and averaged producing a score out of five. This value is then transformed to a score out of 100 by subtracting one and multiplying by 25. The overall DASH score ranged between 0-100. A higher score indicated greater disability.
Time Frame: two week post-surgery compared with six weeks post-surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intramedullary Radius Fixation (Micronail) - Group 1 | Volar Plate Fixation - Group 2
Number analyzed (Participants) | 30 | 30
units on a scale | 24.6 (3.0) | 26.8 (3.1)

ADVERSE EVENTS:
Arm/Group | Intramedullary Radius Fixation (Micronail) - Group 1 | Volar Plate Fixation - Group 2
All-Cause Mortality (participants affected / at risk) | 2/30 | 1/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 3/30 | 2/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intramedullary Radius Fixation (Micronail) - Group 1 (N=30) | Volar Plate Fixation - Group 2 (N=30)
Anticipated (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Change in treatment due to observations during surgery
Anticipated (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) — Loss of fracture reduction
Anticipated (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Stiffness requiring removal of hardware
Unanticipated (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Sustained a median nerve contusion from initial injury and required carpal tunnel release three months after fracture fixation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No